CLINICAL TRIAL: NCT04790266
Title: Early Detection of Cardiotoxicity From Systemic and Radiation Therapy in Breast Cancer Patients
Acronym: CARDIOTOX
Status: Completed | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Collaborators: Cardiocentro Ticino (Other); North Estonia Medical Centre (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01395CE3508
Record Dates: First submitted 2021-02-23; First posted 2021-03-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — cCardiac MRI, ecocardiography and cardiotoxicity blood tests will be repeated as previously scheduled
  Other Names: Echocardiography; Cardiotoxicity laboratory tests (troponin, Pro-BNP, hsCRP)

SUMMARY:
To assess the role of myocardial oedema on CMR (T2 mapping) after radiation therapy and cardiotoxic systemic therapy in predicting the incidence of cardiotoxicity, defined as by consensus guidelines* (decline of LVEF ≥10% points with a final LVEF <53%) measured on CMR and ECHO over the time window of 12 months from the end of radiation therapy.

DETAILED DESCRIPTION:
Overall study schedule The Overall Study Schedule is summarized in the assessment schedule (appendix 1).

This study is composed of three subsequent phases: a Run-In Phase, a RT/Systemic Therapy Phase, a Follow-Up Phase.

Run-In Phase The Run-In Phase starts with the first visit (before any cancer treatment), when Screening/Enrollment procedure is performed. This phase will start once a patient has provided WIC to participate in the study and ends the day of treatment start.

Screening / Enrolment Visit Visit will be performed before the expected starting date of treatment.

After a WIC has been obtained from the patient, the patient will be visited by the Investigators and the following information will be gathered:

* Demographic Data (age, height, weight, BMI);
* Medical history (previous and concomitant diseases, previous therapies, family history of CVD);
* Concomitant Medication;
* Physical examination & overall health assessment (including vital signs).
* Pregnancy test (pre- and perimenopausal women). The inclusion and exclusion criteria will be checked and, if the patient complies with all the Inclusion and Exclusion criteria, she will be enrolled into the study

A baseline assessment will be performed by the Investigator:

CMR, ECG and ECHO will be done at the participating centers The patient will be assigned to specific treatment (chemo/immunotherapy and adjuvant radiation therapy +/- aromatase inhibitor/tamoxifen/LhRh agonist). A standard of care treatment will be administered.

Radiotherapy/Systemic therapy Treatment Phase (specific Visit descriptions) SYSTEMIC TREATMENT Blood sample will be scheduled before and, if possible, 24 hours after chemotherapy administration.

* Patients treated with antracyclines regimens will be checked with ECG and ECHO at the end of treatment.
* Blood sample will be scheduled before Trastuzumab administration every three weeks and ECHO will be done after every 4 cycles (3 months).

RADIOTHERAPY For Technical details see appendix 3. Before starting RT patients will be checked clinically the first day of treatment and baseline tests will be done.

Biomarkers will be checked the first day and in the middle of RT. If a patient gets symptomatic heart failure during the treatment, or if LVEF decline greater than 10% points with a final LVEF <53% measured on Echo, the patient will be referred to the cardiologist for a specific treatment as described by guidelines

End of RT Group Patients treated with trastuzumab, will continue the treatment up to 1 year. Blood tests will be taken every three weeks and Echos will be done after every 4 cycles (3-week cycles).

Follow-Up Phase 2 weeks+/-3 days after the end of RT, blood sample will be taken. An ECHO and CMR will be done.

All patients will be checked 6 weeks after the end of radiotherapy for the study visit.

The following activities will be performed:

Blood sample for biomarkers. If hs-CRP ≥3mg/l, ECHO will be done. All patients will be followed at least until 10 years after the end of RT. Blood samples for measuring biomarkers and ECHO and CMR will be done 12 months after the end of RT.

Unscheduled Visit An unscheduled visit may occur at any time during the study, only for safety reason or for a premature discontinuation from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed
2. Age ≥ 18 years at visit 1
3. Performance status ECOG 0-1
4. *Stage I-III histology proven breast cancer
5. Treated with adjuvant radiotherapy and neo/adjuvant anthracycline and/or trastuzumab-based therapy +/- hormonal therapy
6. Negative pregnancy test (plasma HCG) for all females of childbearing potential (i.e not permanently sterilised- post hysterectomy or tubal ligation status) In the ancillary study patients with stage 0 (DCIS) histology proven breast cancer will also be included.

Exclusion Criteria:

1. Known metastatic spread of any cancer
2. Known active or recurrent hepatic disorder (cirrhosis, hepatitis), ASAT/ALAT 2xULN
3. Renal function decrease (eGFR < 30 ml/min)
4. Known coronary artery disease
5. Angina pectoris
6. Positive or missing pregnancy test (pre- and perimenopausal women) at enrolment visit
7. Patients with baseline LVEF <53% and GLS <15%
8. Patients with pacemaker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged ≥ 18 years with stage I-III breast cancer treated with radiation therapy and neo/adjuvant chemo/immunotherapy +/- aromatase inhibitor/tamoxifen/LhRh agonist.
  An ancillary study will enroll also stage 0 patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
CMR T2 mapping | Time window of 12 months from the end of radiation therapy
  To assess the role of myocardial oedema on CMR (T2 mapping) after radiation therapy and cardiotoxic systemic therapy in predicting the incidence of cardiotoxicity, defined as by consensus guidelines* (decline of LVEF ≥10% points with a final LVEF <53%).

SECONDARY OUTCOMES:
GLS | Time window of 12 months from the end of radiation therapy
  To detect GLS decrease >15% from baseline, measured on Echo over the time window of 12 months
Myocardial edema | Time window of 12 months from the end of radiation therapy
  To assess the incidence of myocardial oedema on CMR (T2 mapping) after radiation therapy and cardiotoxic systemic therapy.
  To assess the incidence of myocardial oedema on ECHO after radiation therapy and cardiotoxic systemic therapy.
Biomarkers (Troponine, pro-BNP, hs-CRP) correlate with LVEF | Time window of 12 months from the end of radiation therapy
  To see if the changes in Troponine (ng/L) will correlate with LVEF measurements, assessed by ECHO. To see if the changes in Troponine (ng/L) will correlate with LVEF measurements, assessed by CMR.
  To see if the changes in pro-BNP (ng/L) will correlate with LVEF measurements, assessed by ECHO.
  To see if the changes in pro-BNP (ng/L) will correlate with LVEF measurements, assessed by CMR.
  To see if the changes in hs-CRP (mg/L) will correlate with LVEF measurements, assessed by ECHO.
  To see if the changes in hs-CRP (mg/L) will correlate with LVEF measurements, assessed by CMR.
Biomarkers (Troponine, pro-BNP, hs-CRP) correlated with GLS | Time window of 12 months from the end of radiation therapy
  To see if the changes in Troponine (ng/L) will correlate with GLS measurements, assessed by ECHO.
  To see if the changes in pro-BNP (ng/L) will correlate with GLS measurements, assessed by ECHO.
  To see if the changes in hs-CRP (mg/L) will correlate with GLS measurements, assessed by ECHO.
Time to biomarkers (Troponine, pro-BNP, hs-CRP) increase | Time window of 12 months from the end of radiation therapy
  To compare the time to the Troponine (ng/L) positivity to the time to the decrease in GLS >15% and/or decline of LVEF ≥10% points with a final LVEF <53% measured on Echo.
  To compare the time to the pro-BNP (ng/L) positivity to the time to the decrease in GLS >15% and/or decline of LVEF ≥10% points with a final LVEF <53% measured on Echo.
  To compare the time to the hs-CRP (mg/L) positivity to the time to the decrease in GLS >15% and/or decline of LVEF ≥10% points with a final LVEF <53% measured on Echo.
Biomarkers (Troponine, pro-BNP, hs-CRP) predictors of cardiotoxicity | Time window of 12 months from the end of radiation therapy
  To see if the changes in Troponine (ng/L) will correlate with developement of cardiotoxicity, defined as by decline of LVEF ≥10% points with a final LVEF <53%.
  To see if the changes in pro-BNP (ng/L) will correlate with developement of cardiotoxicity, defined as by decline of LVEF ≥10% points with a final LVEF <53%.
  To see if the changes in hs-CRP (mg/L) will correlate with developement of cardiotoxicity, defined as by decline of LVEF ≥10% points with a final LVEF <53%.
Major cardiovascular events | follow-up
  To detect major cardiovascular events (defined as acute myocardial infarction, hospitalization due to heart failure, atrial flutter/fibrillation, ventricular tachycardia) or death due cardiac problems during the follow up
cardiac fibrosis | through study completion, an average of 1 year
  assess the role of fibrosis on CMR (T1 mapping with evaluation of extracellular volume) after cardiotoxic radiation therapy and systemic therapy in predicting the incidence of cardiotoxicity
acute asymptomatic pericarditis | through study completion, an average of 1 year
  incidence of acute asymptomatic pericarditis after radiation therapy, measured on CMR
cardiac edema | through study completion, an average of 1 year
  investigate if the area of the edema on CRM correlates with RT dose distribution

CONTACTS AND LOCATIONS:
Overall Officials: mariacarla Valli, Principal Investigator — IOSI
Locations (1):
- Oncology Institute of Italian Switzerland, Bellinzona, Canton Ticino, Switzerland

REFERENCES:
- [Derived] Borgonovo G, Vettus E, Greco A, Leo LA, Faletra FF, Klersy C, Curti M, Valli M. Early Detection of Cardiotoxicity From Systemic and Radiation Therapy in Patients With Breast Cancer: Protocol for a Multi-Institutional Prospective Study. JMIR Res Protoc. 2022 Apr 21;11(4):e31887. doi: 10.2196/31887. PMID 35451989

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT04790266/Prot_SAP_000.pdf